CLINICAL TRIAL: NCT04632043
Title: Effect of Early versUs Delayed intubatiOn on Clinical Outcomes of Patients With COVID-19 (EUDOCO): a Feasibility Randomized Controlled Trial
Brief Title: Early Versus Delayed Intubation of Patients With COVID-19
Acronym: EUDOCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient rate of recruitment
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Ilias Siempos, Pulmonologist, Intensivist, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32635, 13-10-2020
Record Dates: First submitted 2020-11-15; First posted 2020-11-17 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Acute Hypoxemic Respiratory Failure
Keywords: COVID-19
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intubation (Active Comparator): Patients with COVID-19 suffering from severe acute hypoxemic respiratory failure (defined as the need for non-rebreather mask or high flow nasal oxygen with setting FiO2 of at least 90% or non-invasive mechanical ventilation to maintain a SpO2 >92%) for at least 48 hours will undergo intubation.
  Interventions: Other: Endotracheal intubation
- Delayed intubation (Active Comparator): Patients with COVID-19 suffering from severe acute hypoxemic respiratory failure (defined as the need for non-rebreather mask or high flow nasal oxygen with setting FiO2 of at least 90% or non-invasive mechanical ventilation to maintain a SpO2 >92%) for at least 48 hours will continue to receive non-rebreather mask, high-flow nasal oxygen or non-invasive mechanical ventilation in an attempt to avoid intubation.
  Interventions: Other: Endotracheal intubation

INTERVENTIONS:
Other: Endotracheal intubation — Endotracheal intubation

SUMMARY:
Although management of acute hypoxemic respiratory failure associated with coronavirus disease 2019 (COVID-19) often includes mechanical ventilation, the optimal timing of initiation of invasive mechanical ventilation remains unknown.

We hypothesise that a randomized controlled trial comparing early intubation as opposed to delayed intubation among patients with COVID-19 suffering from severe acute hypoxemic respiratory failure is feasible.

DETAILED DESCRIPTION:
A common manifestation of COVID-19 is severe acute hypoxemic respiratory failure. Management of acute hypoxemic respiratory failure associated with COVID-19 often includes mechanical ventilation. The optimal timing of initiation of invasive mechanical ventilation remains unknown.

On the one hand, early initiation of invasive mechanical ventilation (i.e. early endotracheal intubation) has been advocated as a means to reduce subsequent possible aerosolization of the virus, as would happen by alternate means of oxygenation/ventilation allowing air leaks. Also, early intubation may prevent the induction of self-inflicted lung injury in patients who breath spontaneously and have high respiratory drive and, therefore, large transpulmonary pressure swings. On the other hand, delaying intubation, by trying alternate means of oxygenation/ventilation, may mean that some of the patients may not be intubated at all and therefore will be protected from the adverse events of invasive mechanical ventilation (such as ventilator-induced lung injury, ventilator-associated pneumonia and ventilator-induced diaphragmatic dysfunction). The latter strategy may also address the unavailability of enough ventilators to meet the increased demand of treating patients with COVID-19.

Given that no randomized controlled trials are currently available to guide clinical practice regarding optimal timing of intubation, we propose a single-center randomized controlled feasibility trial to compare early intubation versus delayed intubation among patients with COVID-19 suffering from severe acute hypoxemic respiratory failure. The aim is that we gain experience and produce pilot data, which could inform the design of a subsequent large multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with confirmed COVID-19 and severe acute hypoxemic respiratory failure

Exclusion Criteria:

* Postoperative acute respiratory failure (within one week from surgery)
* After cardiac arrest
* Chronic hypoxemic respiratory failure
* Hypercapnic respiratory failure
* No full code
* Lack of equipoise of the clinical team
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Time from onset of severe acute hypoxemic respiratory failure to intubation | 28 days
  Difference in time from onset of severe acute hypoxemic respiratory failure to intubation between the two groups will be the primary (feasibility) outcome

SECONDARY OUTCOMES:
Organ failure-free days | 28 days
  Number of days without the need for invasive mechanical ventilation, vasopressors and continuous renal replacement therapy with days after death not to be considered as organ failure-free days
Need for continuous renal replacement therapy | 28 days
Ventilator-free days | 28 days
ICU-free days | 28 days
  Intensive care unit-free days
Mortality | 28 days
  All-cause ICU-mortality
Number of severe post-intubation adverse events | Within 30 minutes from intubation
  Cardiac arrest and severe arterial desaturation (defined as SpO2 <80% for >5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Ilias Siempos, MD, DSc, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 3 months from publication
Access Criteria: To anyone who is interested in writing a meta-analysis or review.

REFERENCES:
- [Result] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Fan E, Beitler JR, Brochard L, Calfee CS, Ferguson ND, Slutsky AS, Brodie D. COVID-19-associated acute respiratory distress syndrome: is a different approach to management warranted? Lancet Respir Med. 2020 Aug;8(8):816-821. doi: 10.1016/S2213-2600(20)30304-0. Epub 2020 Jul 6. PMID 32645311
- [Result] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Result] Bauer PR, Gajic O, Nanchal R, Kashyap R, Martin-Loeches I, Sakr Y, Jakob SM, Francois B, Wittebole X, Wunderink RG, Vincent JL; ICON Investigators (Supplemental Appendix 1). Association between timing of intubation and outcome in critically ill patients: A secondary analysis of the ICON audit. J Crit Care. 2017 Dec;42:1-5. doi: 10.1016/j.jcrc.2017.06.010. Epub 2017 Jun 16. PMID 28641231
- [Result] Kang BJ, Koh Y, Lim CM, Huh JW, Baek S, Han M, Seo HS, Suh HJ, Seo GJ, Kim EY, Hong SB. Failure of high-flow nasal cannula therapy may delay intubation and increase mortality. Intensive Care Med. 2015 Apr;41(4):623-32. doi: 10.1007/s00134-015-3693-5. Epub 2015 Feb 18. PMID 25691263